CLINICAL TRIAL: NCT03041077
Title: Influence of Instaflex Advanced Supplement on Joint Function: A Randomized, Placebo-controlled Community Trial
Brief Title: Influence of Instaflex Advanced Supplement on Joint Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Direct Digital (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0081
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Knee Discomfort

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instaflex Advanced (Experimental): Dietary supplement: Joint function
  Interventions: Dietary Supplement: Instaflex Advanced
- Placebo (Placebo Comparator): Dietary supplement: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Instaflex Advanced — Joint function
  Arms: Instaflex Advanced
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Joint discomfort is reported by 32% of U.S. adults, and increases with age. The knee is the most common site of joint discomfort regardless of age. Nearly half of people with knee joint discomfort use natural supplements to alleviate symptoms, but more research is needed to determine their effectiveness. In a previous study, we measured the effect of 8-weeks ingestion of a commercialized joint support dietary supplement (InstaflexTM Joint Support, Direct Digital, Charlotte, NC) compared to placebo on joint discomfort, stiffness, and function in adults with self-reported joint discomfort. This study will be repeated using Instaflex Advanced, with a longer 12-week time period. The Instaflex Advanced supplement includes six products: turmeric, resveratrol, Boswellia serrata, collagen, hyaluronic acid, and black pepper extract. This unique blend may improve joint function and increase mobility, but has not yet been tested in humans using a randomized, double-blinded, placebo-controlled research design. The primary purpose of this study is to assess the effect of 12-weeks ingestion of the Instaflex Advanced supplement compared to placebo in improving knee function in adults with self-reported knee joint discomfort.

DETAILED DESCRIPTION:
The research procedures will be conducted at the Human Performance Laboratory (Room 1201, Plants for Human Health Institute Building, 600 Laureate Way), operated by Appalachian State University at the North Carolina Research Campus (NCRC) in Kannapolis, NC. Subjects will come here for orientation/baseline testing and then 3 other lab visits (each session will take about 30 minutes). The total amount of time study participants will be asked to volunteer for this study is about 2 hours at the Human Performance Laboratory (over a 12-week period). Participants will also take a daily supplement for 12 weeks and keep compliant with this regimen.

Lab visit testing sequence:

1. First visit:

   1. Consent form
   2. Medical health questionnaire to verify medical history, and lifestyle habits.
   3. Questionnaire for previous 4-weeks symptoms.
   4. Height, weight, and percent body fat (BIA).Testing will take place behind a screened area of the lab to maintain privacy.
   5. Questionnaires: WOMAC, visual pain scale, POMS.
   6. Receive supplement organizer tray with 4-weeks supply (and instructions).
   7. After a practice trial, study participants will walk as quickly and far as they can on a track for 6 minutes. Total distance covered in 6 minutes will be recorded.
2. 4 weeks, 8-weeks, 12 weeks (second, third, and fourth lab visits):

   1. Symptoms log for previous 4-weeks symptomatology.
   2. Height, weight, and percent body fat.
   3. Questionnaires: WOMAC, visual pain scale, POMS.
   4. Receive supplement organizer tray with 4-weeks supply (and instructions) during second and third lab visits.
   5. 6-minute walk test

Supplements:

Supplements (Instaflex Advanced, placebo) will be contained in identical looking capsules and organized by day of the week in supplement organizer trays. Study participants will take 1 capsule each day in the morning. The placebo capsules contain magnesium stearate, an inert substance. The Instaflex Advanced supplement ingredients include: turmeric, resveratrol, Boswellia serrata, collagen, hyaluronic acid, and black pepper extract. Compliance will be monitored with bi-weekly email messages, and by counting unused capsules when the supplement trays every 4 weeks. Acetaminophen, as found in Tylenol, will be allowed as a rescue medicine for pain during the study as needed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult
* Age 50-75 years
* Self-reported history (>3 months) of joint discomfort in the knees. NOTE: the severity of knee discomfort will be determined through a questionnaire called the WOMAC, and should be at least 2 points (indicating mild knee discomfort or greater).
* No history of regular use of non-steroidal anti-inflammatory drugs (NSAIDs) use (e.g., ibuprofen, aspirin) during the previous two weeks, and willingness to avoid the use of NSAIDs during the 12-week study.
* Not on other medications (e.g., analgesic gels, arthritis medications, other anti-inflammatory drugs) or supplements (in particular, glucosamine and chondroitin) for joint discomfort during the previous two weeks, and a willingness to avoid use of these during the 12-week study.
* No serious medical problems (current cancer case, severe rheumatoid arthritis, recent heart attack, recent stroke, congestive heart failure, ulcers, kidney disease, or other disease that would interfere with study participation).
* No psychiatric disorder or other condition that might interfere with self-assessment ability.
* Willingness to follow all study procedures including randomization to one of two groups, and to stay weight stable during the study.

Exclusion Criteria:

* Inability to comply with study requirements including avoidance of NSAIDs, other anti-inflammatory medications, or discomfort supplements.
* Current diagnosis of cardiovascular disease, cancer (except for non-melanoma skin cancer), severe rheumatoid arthritis, ulcers, kidney disease, psychiatric disorder.
* For female subjects: Pregnant or nursing, or planning to be pregnant or nursing during the study.
* On a weight loss program during the study.
* Vegetarian or vegan.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported on questionnaire
Enrollment: 66 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC total score | Change from baseline WOMAC total score at 4 weeks, 8 weeks, 12 weeks
  WOMAC questionnaire responses pre-study, 4 weeks, 8 weeks, 12 weeks

SECONDARY OUTCOMES:
WOMAC subscales of pain, stiffness, and physical function | Change from baseline WOMAC subscales at 4 weeks, 8 weeks, 12 weeks
  WOMAC questionnaire subscale responses pre-study, 4 weeks, 8 weeks, 12 weeks
Visual Pain Scale | Change from baseline visual pain scale at 4 weeks, 8 weeks, 12 weeks
  10-point Likert-type scale for knee pain severity
Profile of Mood States (POMS) | Change from baseline POMS at 4 weeks, 8 weeks, 12 weeks
  Assessment of mood state
6 minute Walk Test | Change from baseline 6 minute walk test at 4 weeks, 8 weeks, 12 weeks
  Maximum distance covered during 6 minutes of walking

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan